CLINICAL TRIAL: NCT06247449
Title: MRI Screening for Brain Metastases Among Patients With Triple Negative or HER2+ Stage II or III Breast Cancer: A Multi-centre Prospective Cohort Study
Brief Title: MRI Screening for Brain Metastases Among Patients With Triple Negative or HER2+ Stage II or III Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Princess Margaret Hospital, Canada (Other); MOUNT SINAI HOSPITAL (Other); Trillium Health Partners (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SUN#5967
Record Dates: First submitted 2024-01-25; First posted 2024-02-07 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: HER2; Triple Negative; Brain Metastasis
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — Neuroimaging

STUDY DESIGN:
Intervention Model Description: Patients (30 with TN and 30 with HER2+ breast cancer) will be recruited initially as part of a 2-stage design. If at least 1 out of 30 recruited patients is diagnosed with a BrM (3.3% incidence), then an additional 70 patients will be recruited to characterize the risk of BrM among 100 patients in the relevant subgroup (TN and/or HER2+).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening MRI (Experimental): One-time contrast-enhanced brain magnetic resonance imaging (MRI), blood draw for circulating tumor DNA and assessment via the Testing Morbidity Index (TMI)
  Interventions: Diagnostic Test: Brain imaging; Diagnostic Test: Analysis of circulating tumor DNA; Behavioral: Testing Morbidities Index

INTERVENTIONS:
Diagnostic Test: Brain imaging — Contrast-enahanced Brain Magnetic Resonance Imaging (MRI)
Diagnostic Test: Analysis of circulating tumor DNA — Blood draw for analysis of circulating tumor DNA
Behavioral: Testing Morbidities Index — Questionnaire regarding the participant's perception of brain imaging.

SUMMARY:
The goal of this multi-centre, prospective study is to assess the frequency of asymptomatic brain metastasis in patients with stage IIb or III Triple Negative or HER2 positive breast cancer. The main questions it aims to answer are:

1. What proportion of patients with stage IIb or III Triple Negative or HER2 positive breast cancer have asymptomatic brain metastases identified on a screening contrast-enhanced magnetic resonance imaging (MRI) of the brain?
2. How do patients feel about undergoing brain imaging to screen for asymptomatic brain metastasis?
3. What clinical as well as liquid and tissue-based biomarkers are associated with asymptomatic detection of brain metastasis?

Participants will undergo brain imaging, provide one blood sample (for analysis of ctDNA), and complete the Testing Morbidities Index (TMI) questionnaire after imaging is done. Procedures may take place either prior to or after completion of (neo)-adjuvant systemic therapy; however, the study interventions must take place within 18 months of initial breast cancer diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18.
2. Triple Negative OR HER2+ breast cancer (as per 2018 ASCO/CAP guidelines).
3. Stage IIb or III disease.
4. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen may participate.
5. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Creatinine clearance <30 mL/min using the Cockcroft-Gault equation (in accordance with the product monograph for Gadavist IV contrast.
2. Pregnant women are not permitted to participate given that the safety of IV contrast is unknown in this population.
3. Patients with central nervous system symptoms that are concerning for brain metastases that would otherwise be referred for brain imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Asymptomatic brain metastasis frequency among HER2+ patients | 18 months
  Proportion of eligible patients with Stage IIb or III HER2+ breast cancer who have asymptomatic brain metastasis
Asymptomatic brain metastasis frequency among Triple Negative patients | 18 months
  Proportion of eligible patients with Stage IIb or III Triple Negative breast cancer who have asymptomatic brain metastasis

SECONDARY OUTCOMES:
Acceptability of brain imaging to patients | 18 months
  Proportion of patients who are approached about the study who agree to enroll
Patients' acceptability of the brain magnetic resonance imaging | 18 months
  Patients' acceptability of the brain magnetic resonance imaging as evaluated by the "Testing Morbidities Index" (TMI)
Proportion of patients who have subsequent brain magnetic resonance imaging | 36 months
  Annual chart review to determine the frequency of patients who have subsequent brain imaging performed after the first trial magnetic resonance imaging

OTHER OUTCOMES:
Exploratory biomarkers | 36 months.
  Evaluate a possible correlation between the presence of circulating tumor DNA in the blood of patients at the time of study enrollment and future development of brain metastases when the study has been completed.
Correlation between circulating tumor DNA in the blood at enrollment and incidence of brain metastases at the end of the study | 36 months.
  Evaluate a possible correlation between the presence of circulating tumor DNA in the blood of patients at the time of study enrollment and the incidence of brain metastases when the study has been completed.

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Jerzak, MD, M.Sc, Principal Investigator — Sunnybrook Health Science Centre
Locations (1):
- Sunnybrook Health Science Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No